CLINICAL TRIAL: NCT03279926
Title: Preschoolers Learning and Active in PlaY
Acronym: PLAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pooja Tandon, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000628; 1R21CA218592-01 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLAY (Experimental): Preschoolers & their teachers will get activity trackers and the child care program/providers will get some basic information on the use of the trackers and how to integrate their use in the curriculum. A PLAY Champion will be identified to help support PLAY related activities.
  Interventions: Behavioral: PLAY
- PLAY Parents (Experimental): Everything in Arm 1 plus one parent per child will receive an activity tracker and will get reports to help with physical activity goal setting for the family.
  Interventions: Behavioral: PLAY; Behavioral: PLAY Parents
- PLAY Teachers (Experimental): Everything in Arm 1 plus an enhanced focus on teacher wellness, specifically with regard to active lifestyles for them.
  Interventions: Behavioral: PLAY; Behavioral: PLAY Teachers

INTERVENTIONS:
Behavioral: PLAY — Activity trackers + curriculum information
Behavioral: PLAY Parents — Enhanced parental engagement
  Arms: PLAY Parents
Behavioral: PLAY Teachers — Enhanced teacher engagement with active living initiates for the teachers
  Arms: PLAY Teachers

SUMMARY:
The overall aim of this proposal is to develop and test early childhood education setting-based physical activity (PA) interventions that are innovative by using wearable technology to facilitate monitoring, feedback and motivation for physical activity across multiple levels (child, parent, educator). We posit that our intervention strategies will promote behavior changes in parents and educators, leading to greater awareness and communication about physical activity, more active play opportunities, and ultimately more physical activity for preschoolers. In the R21, we will test the acceptability, feasibility and initial efficacy of three 6 month early childhood education setting- based, multi-level interventions to promote preschoolers' PA using wearable technology and additional behavior change techniques to engage educators and parents. The results of this study will inform a larger intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* attends preschool in a child care center participating in this study
* no physical/health restrictions on participating in physical activities

Exclusion Criteria:

* unable to participate in all physical activities

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Post-intervention physical activity (children) | Month 6 compared to baseline
  accelerometer measured
Post-intervention physical activity (children) | Month 1 compared to baseline
  accelerometer measured

SECONDARY OUTCOMES:
Active play opportunities at child care | Month 6 compared to baseline
  Using an observation tool, a trained research assistant will note opportunities for active play (including teacher led, child-initiated, outdoor and indoor)

OTHER OUTCOMES:
activity tracker wear | Month 1
  amount of days activity tracker is worn by participant
activity tracker wear | Month 6
  amount of days the activity tracker is worn by participant

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Tandon, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States